CLINICAL TRIAL: NCT05579236
Title: An Observational Longitudinal Cohort Study to Investigate Cortical Disarray Measurement in Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Cortical Disarray Measurement in Mild Cognitive Impairment and Alzheimer's Disease
Acronym: CONGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); Oxford Brain Diagnostics Ltd (Unknown); Cardiff and Vale University Health Board (Other Government); Cardiff University (Other); University of Oxford (Other); Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: RHM NEU0402; NIHR202146 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2022-09-16; First posted 2022-10-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Dementia
Keywords: Neurodegenerative Diseases; Diagnosis; Prognosis; Diagnostic Imaging; Neuroimaging; Magnetic Resonance Imaging; Diffusion Tensor Imaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Neurodegenerative Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants recruited will be invited to join a biosample repository substudy. This is an optional component to the main study that involves the collection and storage of biosamples for analysis of potential biomarkers of Alzheimer's disease and neurodegeneration, to aid validation of the CDM technique, and for future health research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Participants: Patient participants will have a diagnosis of mild cognitive impairment or prodromal / mild Alzheimer's Disease. Participants with a global CDR score of 0.5 and 1 will be recruited in a minimum of a 2:1 ratio respectively in the study.
- Study Companions: Study companions will have sufficient knowledge on the patient participant's condition to complete companion assessments of the patient, in the investigator's judgement, for example they may be carers of the patients.

SUMMARY:
The aim of this study is to find out whether a new image analysis technique called Cortical Disarray Measurement (CDM) could be used to help better diagnose Alzheimer's disease. This study will see whether changes on CDM can be used to identify Alzheimer's disease from a group of people living with memory and thinking problems. The study will also explore how CDM relates to changes in memory or thinking over time.

DETAILED DESCRIPTION:
This is a multi-centre observational longitudinal cohort study to evaluate and optimise the Cortical Disarray Measurement (CDM) technique for diagnosis and prognosis in patients with mild cognitive impairment and prodromal / mild Alzheimer's Disease. CDM is a novel MRI analysis tool that quantifies cortical and regional diffusion tensor imaging signals in grey matter to observe pathological changes related to neurodegeneration. Participants in this study will be monitored for 2 years.

Research Aims:

* Assess the accuracy of CDM in detecting progressive change in cognitive and functional measures over 2 years in participants presenting with mild cognitive impairment or early dementia.
* Determine the relationship between CDM (both cross-sectionally and longitudinally) and change on standard cognitive and functional assessment measures.
* Explore patient and companion views and experiences of the diagnostic journey for dementia and their views on CDM implementation.
* To explore the costs and consequences of introducing CDM-augmented MRI as a form of early diagnosis of Alzheimer's disease in people presenting with MCI or mild AD compared to current practice.

ELIGIBILITY:
PATIENT PARTICIPANTS

Inclusion Criteria:

* Diagnosis of mild cognitive impairment (MCI) or prodromal Alzheimer's Disease (AD) as defined by National Institute on Ageing/Alzheimer's Association (NIA/AA) diagnostic criteria for MCI/prodromal AD, NOT including MCI unlikely due to AD; OR, Diagnosis of Alzheimer's disease as defined by NIA/AA criteria for probable AD
* Clinical dementia rating (CDR) scale global score of very mild or mild (0.5 or 1) impairment
* Ability to undergo and tolerate MRI scans, with no contraindications to MRI
* Ability to tolerate blood draws
* Ability to give informed consent to participate in the study

Exclusion Criteria:

* Do not meet the inclusion criteria
* No study companion available
* Individuals with a non-progressive learning disability
* Pregnant or intending to become pregnant during the study

COMPANION PARTICIPANTS

Inclusion Criteria:

* Aged over 18 years
* Sufficient knowledge on study participant's condition to complete companion assessments of the patient, in the investigator's judgement
* Able and willing to attend all clinical visits for completion of companion assessments or provide the relevant assessments remotely via phone or video call

Exclusion Criteria:

* A condition or reason, in the investigator's judgement, that would question the validity of the acquired companion reported data
* Individuals who are not fluent in English

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 200 patient participants and 200 study companions will be recruited to the study. Patient participants will have a diagnosis of mild cognitive impairment or prodromal / mild Alzheimer's Disease. Participants with a global CDR score of 0.5 and 1 will be recruited in a minimum of a 2:1 ratio respectively in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
CDR Progression | Baseline (Study day 1) to month 24
  CDR Progression defined as a binary variable (yes/no) indicating either an increase in global outcome on Clinical Dementia Rating (CDR) scale (which takes value 0, 0.5, 1, 2 or 3, with higher scores reflecting more severe dementia), or an increase greater than, or equal to, 2 points on CDR Sum of Boxes (which takes values from 0 to 18 with higher values indicating a worse outcome)

SECONDARY OUTCOMES:
CDR Sum of Boxes | Baseline (Study day 1) to month 24
  Change from baseline in the Clinical Dementia Rating (CDR) Sum of Boxes. CDR Sum of boxes is the sum over 6 domains (memory, orientation, judgment & problem solving, community affairs, home & hobbies, and personal care), each rated on a 5-point scale (0, 0.5, 1, 2, 3), giving a total score that ranges from 0 to 18, with higher values indicating a worse outcome.
ADAS-cog | Baseline (Study day 1) to month 24
  Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-cog). Higher scores for ADAS-Cog represent a worse outcome.
MMSE | Baseline (Study day 1) to month 24
  Change from baseline in Mini Mental State Examination (MMSE). MMSE ranges from 0 to 30, with lower scores representing a worse outcome.
ADCOMS | Baseline (Study day 1) to month 24
  Change from baseline in Alzheimer's disease composite score (ADCOMS). The range of ADCOMS is between 0 and 1.97, with higher scores representing a worse outcome.
RBANS | Baseline (Study day 1) to month 24
  Change from baseline in the RBANS total score. The repeatable battery for the assessment of neuropsychological status (RBANS) is a brief neuropsychological battery. The total score can classify patients as follows: Average/Mild Impairment (standard scores of 70 or above), Moderate Impairment (standard scores from 55 to 69), and Severe Impairment (standard scores <54), such that lower scores indicate a worse outcome.
ADCS-ADL | Baseline (Study day 1) to month 24
  Change from baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Scale (ADCS-ADL). ADCS-ADL
Functional Activities Questionnaire (FAQ) | Baseline (Study day 1) to month 24
  The Functional Activities Questionnaire (FAQ) measures instrumental activities of daily living. Scores range from 0 (independent) to 30 (dependent), with higher scores indicating a worse outcome.
Institutionalisation or POC | Baseline (Study day 1) to month 24
  Institutionalisation in care home or nursing home or implementation of package of care (POC) for dementia. Binary outcome (yes, no), with "yes" indicating a worse outcome.
Death (any cause) | Baseline (Study day 1) to month 24
  Death due to any cause
EQ-5D-5L (Patient Participant) | Baseline (Study day 1) to month 24
  EuroQuol EQ-5D-5L is an instrument to describe and value health on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
EQ-5D-5L (Study Companion) | Baseline (Study day 1) to month 24
  EuroQuol EQ-5D-5L is an instrument to describe and value health on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Zarit Burden Interview | Baseline (Study day 1) to month 24
  The Zarit Burden Interview (ZBI) assesses caregiver perceptions of burden. Higher scores indicate a worse outcome.
Health and social care resource usage | Baseline (Study day 1) to month 24
  Health and social care resource usage questionnaire. Higher values indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kipps, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust; Steven Chance, PhD, Study Chair — Oxford Brain Diagnostics Ltd
Locations (3):
- United Kingdom (3):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Dorset Healthcare University NHS Foundation Trust, Bournemouth
  - Cardiff and Vale University Health Board, Cardiff